CLINICAL TRIAL: NCT04577937
Title: Sleep Patterns in Patients Affected by Lymphangioleiomiomatosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: dr. Stefano Nava (Other)
Responsible Party: Sponsor-Investigator, dr. Stefano Nava, Professor Stefano Nava, MD-FERS, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Organization: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 270/2016/O/Oss/AOUB
Record Dates: First submitted 2020-06-30; First posted 2020-10-08 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Lymphangioleiomyomatosis; Sleep Disorder; Sleep Apnea Syndromes; Hypopnea Syndrome
MeSH Terms: conditions — Lymphangioleiomyomatosis; Sleep Wake Disorders; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: cohort study, pilot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSG in LAM patients (Experimental): Patients affected by LAM underwent whole-night PSG
  Interventions: Diagnostic Test: LAM patients underwent PSG

INTERVENTIONS:
Diagnostic Test: LAM patients underwent PSG — Patients with confirmed diagnosis of LAM underwent a whole-night polysomnography. The presence of either acute or chronic respiratory failure or the use of long-term oxygen therapy are considered exclusion criteria

SUMMARY:
Lymphangioleiomyomatosis (LAM) is a rare and progressive pulmonary disease of unknown etiology that almost exclusively affects women. It is characterised by cystic radiological lung pattern and by the possible presence of angiomyolipomas in other sites or organs. Functionally LAM is associated with airway obstruction or restriction and progressive hypoxemia up to chronic respiratory failure.

There are no studies, so far, which have investigated whether during sleep these patients show changes in the sleep profile and gas exchange and if these changes are related to disease severity. Aim of the study, prospective and pilot, is to evaluate whether the physiological modification of respiratory mechanics during sleep is associated with polysomnographic alterations in LAM.

DETAILED DESCRIPTION:
Lymphangioleiomiomatosis (LAM) is a rare progressive disease that affects primarily lungs with a cystic radiologic pattern and may be associated with angiomiolipomas in the kidneys or in other sites and an increased frequency of meningioma. Patients with sporadic LAM are usually female (incidence around 1/400.000 adult females). LAM associated with tuberous sclerosis may affect male, female and children.

LAM patients are functionally characterized by obstructive or restrictive syndrome that leads patients to hypoxemia and chronic respiratory failure, so that quality of Life (QoL) of these patients is affected by dyspnea. Hypoxemia contributes to the development of secondary pulmonary hypertension (PH) during progression of LAM history, worsening the damage.

The modifications in the neural control of ventilation during sleep in combination with anatomical disposition drive to sleep-related changes in upper airway resistance and physiologic desaturations. In healthy subjects these features are almost completely compensated but, in LAM patients, may lead to airway obstruction and/or pathologic oxygen desaturation that could be managed. So far, none have investigated the changes in sleep architecture and related blood gas exchange in patients with LAM relating these changes with disease severity.

This pilot study investigate if the physiologic modifications of breathing during sleep lead to sleep disorders in LAM patients, measured through abnormalities in polysomnography (PSG) and ih sleep disorders in LAM are associated with respiratory functional abnormalities and disease severity.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of LAM according to current guidelines
* sign of informed consent to participate

Exclusion Criteria:

* the presence of either acute or chronic respiratory failure
* the use of long-term oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-07-08 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of sleep disorders in LAM | 1 year
  Aim of the project is to assess the presence of sleep disorders (oxygen destaruration during sleep and/or sleep apnea or hypopnea) in patients affected by LAM.
correlation between sleep-related disorders and LAM severity measured by spirometry | 1 year
  Another aim of the project is to stratify the presence of sleep-related disorders (oxygen desaturation during sleep, sleep apnea or hypopnea) according to the severity of LAM measured through functional impairment. By spirometry performed at the time of PSG the study population will be divided in: subjects with obstructive impairment; subjects with restrictive abnormality and subjects with no alterations.
correlation between sleep-related disorders and LAM severity measured by annual decline of forced-expiratory volume at the first second (FEV1) | 1 year
  Another aim of the project is to stratify the presence of sleep-related disorders (oxygen desaturation during sleep, sleep apnea or hypopnea) according to the severity of LAM measured by annual decline of forced-expiratory volume at the first second (FEV1), expressed in ml/year. Annual decline of FEV1 will be measured subtracting the FEV1 value (ml) at the time of PSG test to the FEV1 value (ml) at the time of diagnosis and then, dividing it by disease duration in years.
correlation between sleep-related disorders and LAM severity measured by arterial blood gas exchange | 1 year
  Another aim of the project is to stratify the presence of sleep-related disorders (oxygen desaturation during sleep, sleep apnea or hypopnea) according to the severity of LAM measured through arterial blood gas exchanges values: partial pressure of oxygen (PaO2 - mmHg), partial pressure of carbon dioxide (PaCO2 - mmHg), oxygen saturation (SatO2, %).
correlation between sleep-related disorders and clincal parameters | 1 year
  Moreover, another aim is to assess the distribution of sleep disorders (oxygen desaturation during sleep, sleep apnea or hypopnea) according to age, sex, body mass index (BMI), comorbidities in patients affected by LAM.
  BMI will be calculated using height (mt) and weight (Kg) at the time of PSG and expressed in Kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nava, MD-FERS, Principal Investigator — AOSP - Azienda Ospedaliero Universitaria Di Bologna
Locations (1):
- Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No